CLINICAL TRIAL: NCT01567956
Title: Phase III Randomized Multicenter International Study to Investigate the Safety and Efficacy of Propionyl-L-Carnitine Hydrochloride Modified Release Tablets in Patients Affected by Mild Ulcerative Colitis Under Oral Stable Treatment
Brief Title: Propionyl-L-Carnitine Hydrochloride in Patients With Mild Ulcerative Colitis; Efficacy, Safety and Tolerability Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Evidence of very low probability to success. No safety issues
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST261DM11006; 2011-004770-28 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2014-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propionyl-L-Carnitine (Experimental): Modified release tablets containing 500 mg of propionyl-L-carnitine
  Interventions: Drug: Propionyl-L-Carnitine
- Placebo (Placebo Comparator): Modified release tablets containing inert substances
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propionyl-L-Carnitine — 500 mg modified release tablets, 500 mg bid; treatment duration 8 weeks
  Arms: Propionyl-L-Carnitine
Drug: Placebo — 500 mg inert substances modified release tablets, 500 mg bid; treatment duration 8 weeks
  Arms: Placebo

SUMMARY:
The aim of the trial is to test safety, tolerability and efficacy of Propionyl-L-carnitine modified release tablets 1g/die in reducing the symptoms of the disease with respect to the proportion of patients with disease remission at the end of the 8 weeks of treatment. It will also aim to investigate capability of the treatment in the maintenance of remission after four weeks of treatment interruption; histological changes will be also evaluated and finally, improvement in the overall quality of life as measured by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ) will be investigated.

DETAILED DESCRIPTION:
Although it seems clear that an abnormal function of the colonic epithelium is the central problem causing inflammation and the unusual immunological response to the normal gut flora in inflammatory bowel disease (IBD), the actual causes of these dysfunctions are still unknown. Short Chain Fatty Acids (SCFA) are the main fuel of the colonic epithelium, and are normally produced by the bacterial flora by fermentation of the complex carbohydrates forming non soluble fibers usually introduced with everyday diet. Butyrate alone contributes 70% of the normal colonocyte energy. Studies done using animal models and colonic mucosa biopsies from patients suffering form ulcerative colitis (UC) have consistently shown that a metabolic change occurs in diseased colonic mucosa, with an impairment of butyrate oxidation (and of beta-oxidation) and an energy shortage that is only incompletely compensated by oxidation of glucose and other substrates such as glutamine. It is also well known that matrix metalloproteases production is highly increased in IBD and that serum transglutaminase activity is significantly reduced in patients with IBD. Transglutaminases are enzymes contributing to the crosslinking of matrix proteins and the reduction seen in patients affected by IBD correlates well with the endoscopic and histopathologic grading in UC, meaning that part of the circulating enzyme is sequestered in the injured colonic tissue in the effort to re-build the extracellular matrix during the healing process. Propionyl-L-carnitine Hydrochloride (PLC) is a molecule that has already been shown to reduce membrane lipid peroxidation in endothelial cells from bovine aorta and coronary vessels, to reduce the effects of hypoxia in coronary endothelial cells, and to play a role in the cardiac metabolic abnormalities that contribute to the mechanical dysfunctions leading to heart failure. Given these properties of Propionyl-L-carnitine Hydrochloride (ST 261) and given the peroxidative damage suffered by colonocytes in UC together with their metabolic impairment, the use of this molecule for the treatment of UC seemed to be appropriate and sound, in particular as a carrier of a propionate moiety that, once transformed into succinate, enters the Kreb cycle, acting as an extra burst fuel improving the balance of energy production inside tissues. Previous clinical experience has shown that PLC promoted complete or nearly complete regression of cutaneous trophic ulcers in a large number of vasculopathic patients refractory to all other therapies. As far as the UC pathology is concerned, the effects of ST 261, given orally or intrarectally, were investigated at different dosages, in preclinical experimentation, either after a single trinitrobenzene sulphonic acid (TNBS) administration (acute colitis) or after repeated TNBS administrations (reactivated colitis). The results showed a reduction in the damaged colon area both in acute model and reactivated colitis, even if the beneficial effect of restoration of TNBS-induced alterations of tissue morphology is more evident in the reactivated colitis model, particularly after oral administration. Based on the above-described results a development plan in humans started to investigate the activity of PLC in the treatment of ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Have read the Information for the Patient and signed the Informed Consent Form.
* Diagnosis of active ulcerative colitis since at least 4 weeks as confirmed endoscopically and histologically.
* Disease Activity Index comprised between 3 and 6, inclusive (mild ulcerative colitis), with rectal bleeding sub-score of at least 1.
* Stable background oral aminosalicylates (mesalazine, balsalazide, olsalazine) or sulfasalazine standard therapy for greater than or equal to 4 weeks prior to screening assessments.
* If female, not pregnant or nursing. For women of childbearing potential, willingness to avoid a pregnancy during the treatment period and for at least 4 weeks from the last dose of drug and utilization of an efficient method of birth control for the entire duration of the trial and until the first menses after a 30-day period after the last dose of trial medication.

Exclusion Criteria:

* Crohn's disease and indeterminate colitis.
* Current or previous (in the last 10 days preceding the screening) use of systemic corticosteroids.
* Use of systemic antibiotics in the last 10 days preceding the screening.
* Use of systemic Nonsteroidal anti-inflammatory drugs on a repeat basis in the last 10 days preceding the screening.
* Use of probiotics started within 10 days preceding the screening. A stable regimen from at least 10 days prior to screening is allowed but the patient must be willing to continue up to the end of the study.
* Use of immunosuppressants or biological agents within the last 6 weeks preceding the screening.
* Treatment with L-carnitine or its esters derivatives within the last 3 months.
* Stool culture positive for enteric pathogens (eg, Shigella, Salmonella, Yersinia, Campylobacter) or toxins (C.difficile).
* Significantly impaired liver, renal, pulmonary or cardiovascular function as assessed by the investigator.
* History of colon resection.
* Diverticulitis, symptomatic diverticulosis.
* Active peptic ulcer disease.
* Proctitis (extent of inflammation < 15 cm from the anus).
* Bleeding disorders
* Rectal therapy with any therapeutic enemas or suppositories with the exception of those required for endoscopy during the 10 days preceding the screening.
* Active or chronic infection(s) or malignancies.
* Known hypersensitivity to the active ingredient and excipients of the study drug
* Patients treated with L-Carnitine or its esters derivatives during the 3 months preceding the screening phase.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Proportion of clinical/endoscopic remissions | End of treatment (week 8)
  Remission will be defined according with the overall modified Mayo score (Disease Activity Index). A score ≤ 2 with rectal bleeding sub-score = 0 and no other individual sub-score >1 will be considered necessary to classify the patient in remission state.

SECONDARY OUTCOMES:
Change from baseline in Rectal bleeding evaluation | At week 2, 6 and 8 of treatment and after 4 week follow-up
  Evaluation will be performed by means of Disease Activity Index (DAI) sub-score (from 0 to 3).
Change from baseline in stool frequency evaluation | At week 2, 6 and 8 of treatment and after 4 week follow-up
  Evaluations will be performed by means of Disease Activity Index (DAI) sub-score (from 0 to 3).
Histological response to the treatment | End of treatment (week 8)
  Evaluated as an improvement of the histological index of at least 1 point
Change from baseline in C-reactive protein (CRP) and Fibrinogen | End of the treatment (week 8) and after 4 week follow-up
Improvement of patients quality of life | End of treatment period (week8) and after 4 week follow-up
  A validated specific questionnaire, the SIBDQ by McMaster university will be administered to evaluate changes in patients' quality of life
Haematology | Baseline and end of treatment (week8)
  Haemoglobin, Haematocrit, RBC, WBC and differential count.
Electrocardiogram | At baseline and at the end of treatment period (week8)
  Standard intervals (PR, RR, QRS, QT) will be collected plus all rhythm abnormalities
Adverse Events collection | 12 weeks
Serum Chemistry | At baseline and at the end of treatment period (week8)
  Standard evaluation including renal and liver function, electrolytes and blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Ardizzone, MD, Study Chair — Head of Inflammatory Bowel Diseases Unit Hospital "Luigi Sacco" Milan - ITALY
Locations (58):
- Austria (4):
  - Landeskrankenhaus-Universitätskliniken Innsbruck - Klinische Abteilung für Gastroenterologie und Hepatologie, Innsbruck
  - Krankenhaus der Barmherzigen Brüder - Abteilung für Innere Medizin, Salzburg
  - Allgemeines Krankenhaus Wien - Universitätsklinik Klinik für Innere Medizin III, Vienna
  - Ordinationszentrum Döbling, Vienna
- France (9):
  - Centre Hospitalier Intercommunal Créteil 40 avenue de Verdun, Créteil
  - Centre Hospitalier Universitaire Hôpital Nord - Service D'Hépato-Gastro-Entérologie, Marseille
  - Centre Hospitalier Universitaire Hotel Dieu Service d'hépato-gastroentérologie, Nantes
  - Hôpital de I´Archet 2 Service d'Hépato-Gastroentérologie et de Nutrition Clinicque, Pôle Digestif, Nice
  - Hôpital Nord - Dept. of Gastroenterology, Picardie
  - Hôpital Robert Debré Service et Consultation d'Hépato-Gastro-Entérologie, Reims
  - Hopital Nord - CHU de Saint-Etienne Service de Gastro-Entérologie, Saint-Etienne
  - Hôpital Rangueil Service de gastro-enterologie, Toulouse
  - Hôpital Brabois Service de gastro-enterologie, Vandœuvre-lès-Nancy
- Germany (11):
  - Charité Universitätsmedizin Berlin Universitätsklinik Charité, Campus Mitte Medizinische Poliklinik, Berlin
  - Saint Josef Hospital Ruhr Universitaet Bochum Gudrunstraße 56, Bochum
  - Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum Dresden Medizinische Klinik und Poliklinik I, Dresden
  - Universtätsklinikum Schleswig-Holstein Gastroenterologie, Lübeck
  - Universitätsklinikum Magdeburg A.ö.R. Klinik für Gastroenterologie, Hepatologie und Infektiologie, Magdeburg
  - Universitätsmedizin Mannheim II. Medizinische Klinik, Mannheim
  - Praxis Prof. Dr. med. Herbert Kellner, München
  - Universitätklinikum Münster Medizinische Klinik und Poliklinik für Innere Medizin, Münster
  - Gastroenterologische Fachpraxis am Germania Campus, Münster
  - Elbe Klinikum Stade Innere Medizin, Abteilung Gastroenterology, Stade
- Hungary (10):
  - Fovárosi Önkormányzat Péterfy Sándor Utcai Kórház, Budapest
  - Semmelweis Egyetem 1st Internal Dept., Budapest
  - Pannónia Magánorvosi Centrum Kft., Budapest
  - Semmelweis Egyetem II. sz. Belgyógyászati Klinika, Budapest
  - Békés Megyei Képviselotestület Pándy Kálmán Kórháza Semmelweis ulica 1, Gyula
  - Kaposi Mór Megyei Oktató Kórhaz Belgyógyászati Osztály, Kaposvár
  - Borsod Abaúj Zemplén Megyei Kórház és Egyetemi Oktató Kórház II. sz. Belgyógyászati Osztály, Miskolc
  - Karolina Kórház Rendelointézet Belgyógyászat- Gasztroenterológiai Osztály, Mosonmagyaróvar
  - Clinfan Kft. SMO, Szekszárd
  - CRU Hungary Kft., Szikszó
- Latvia (4):
  - Daugavpils Central Regional Hospital, Daugavpils
  - Paula Stradina Clinical University Hospital Gastroenterology Centre, Riga
  - Latvian Maritime Medicine Centre, Riga
  - Digestive Disease Center GASTRO, Riga
- Lithuania (4):
  - Lietuvos sveikatos mokslu universiteto ligonine VšI Kauno klinikos Gastroenterologijos skyrius, Kaunas
  - Klaipedos jurininku ligonine Diagnostikos skyrius, Klaipėda
  - VšI Mykolo Marcinkeviciaus ligonines, Vilnius
  - Vilniaus universiteto ligonine Santariškiu klinikos Hepatologijos, gastroenterologijos ir dietologijos centras, Vilnius
- Poland (9):
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp.J, Ksawerów
  - SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego Oddzial Gastroenterologii Ogólnej i Onkologicznej, Lódz
  - Wojewódzki Szpital Specjalistyczny w Olsztynie Oddzial Gastroenterologii, Olsztyn
  - Endoskopia Sp. z o.o., Sopot
  - Nzoz Vivamed, Warsaw
  - Akademicki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu Klinika Gastroenterologii i Hepatologii, Wroclaw
  - Wojewodzki Szpital Specjalistyczny im. J. Gromkowskiego we Wroclawiu Oddzial Gastroenterologii, Wroclaw
  - LexMedica, Wroclaw
  - ARS MEDICA s.c., Rybak Maria, Rybak Zbigniew, Wroclaw
- Spain (7):
  - Fundación Hospital de Alcorcón Servicio de Gastroenterología, Alcorcón
  - Centro Medico Teknon Servicio de Aparato Disgestivo, Barcelona
  - Hospital Universitario Virgen de la Arrixaca Servicio de Digestivo, El Palmar
  - Hospital Universitario La Princesa Unidad de Hepatología, Servicio de Gastroenterologia, Madrid
  - Hospital Universitario La Paz Servico de Gastroenterologia, Madrid
  - Corporació Sanitaria Parc Taulí Servicio de Digestivo, Sabadell
  - Hospital Universitario Marques de Valdecilla Servicio de Digestivo, Santander

IPD SHARING:
Plan to Share IPD: No